CLINICAL TRIAL: NCT01747668
Title: Impact of Nutrient Supplementation on Breast Milk Levels of Lactating Women
Brief Title: Lactation Fortification Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL05
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Lactation
Keywords: Mother and Infant Pairs
MeSH Terms: conditions — Breast Feeding | interventions — Soybean Oil; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Supplement (Placebo Comparator): soft-gel placebo capsules, 2 capsules from the placebo bottle per day
  Interventions: Dietary Supplement: Placebo (soybean oil and dl-alpha-tocopheryl acetate)
- Experimental Supplement A (Experimental): soft-gel capsules; 1 capsule from the experimental bottle and 1 capsule from the placebo bottle per day
  Interventions: Dietary Supplement: Similac Prenatal Vitamin soft-gel capsule; Dietary Supplement: Placebo (soybean oil and dl-alpha-tocopheryl acetate)
- Experimental Supplement B (Experimental): soft-gel capsules; 2 capsules from the experimental bottle per day
  Interventions: Dietary Supplement: Similac Prenatal Vitamin soft-gel capsule

INTERVENTIONS:
Dietary Supplement: Similac Prenatal Vitamin soft-gel capsule — One capsule per day for Experimental Supplement A Group; Two capsules per day for Experimental Supplement B Group
  Arms: Experimental Supplement A; Experimental Supplement B
Dietary Supplement: Placebo (soybean oil and dl-alpha-tocopheryl acetate) — Two capsules per day for the Placebo Group; One capsule per day for the Experimental Group A
  Arms: Control Supplement; Experimental Supplement A

SUMMARY:
To investigate the impact of nutrient supplementation during lactation on levels in breast milk.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for the study if they meet all of the following inclusion criteria:

1. Mother with singleton birth, 37-42 weeks gestation and ≥ 2490g
2. Pre-pregnancy BMI </= 30
3. Mother is ≥ 18 years of age
4. Mother is 4-6 weeks postpartum and has been successfully continuously lactating
5. Mother agrees to abstain from the use of any Docosahexaenoic acid (DHA), lutein and/or vitamin E containing supplements for at least 10 days prior to providing a baseline breast milk sample
6. Mother agrees to abstain from the use of non-study supplements throughout the study
7. Mother plans to continue breastfeeding for at least 6 weeks from the start of the study
8. No significant ongoing medical problems in the infant as determined from infant's medical history as related by the parent(s) to the enrolling center personnel

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

1. Subject had adverse maternal and/or fetal medical history
2. Subject is participating in a non-Abbott approved concomitant trial
3. Mother is taking cholesterol medication and/or medication affecting lipid absorption and/or transport

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Breast milk concentration of carotenoids | 1 - 43 days

SECONDARY OUTCOMES:
Breast milk concentration of fatty acids | 1 - 43 days

OTHER OUTCOMES:
Blood levels of nutrients and fatty acids | 1 and 43 days
  In mothers at 1 and 43 days In infants at 43 days

CONTACTS AND LOCATIONS:
Overall Officials: Christina Sherry, PhD, RD, Study Chair — Abbott Nutrition
Locations (6):
- United States (6):
  - Northpoint Pediatrics, LLC, Indianapolis, Indiana
  - Ohio Pediatric Research Association, Inc, Dayton, Ohio
  - Ohio Pediatric Research Association, Inc, Kettering, Ohio
  - Institute of Clinical Research, Mayfield Heights, Ohio
  - The Cleveland Pediatric Research Center, LLC, Parma, Ohio
  - The Cleveland Pediatric Research Center, LLC, Westlake, Ohio

REFERENCES:
- [Derived] Sherry CL, Oliver JS, Renzi LM, Marriage BJ. Lutein supplementation increases breast milk and plasma lutein concentrations in lactating women and infant plasma concentrations but does not affect other carotenoids. J Nutr. 2014 Aug;144(8):1256-63. doi: 10.3945/jn.114.192914. Epub 2014 Jun 4. PMID 24899160